CLINICAL TRIAL: NCT05514730
Title: Treatment for Problematic Sexual Behavior of Preteen Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Brian Allen, Psy.D., Associate Professor of Pediatrics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00020807
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Problematic Sexual Behavior Among Preteen Children
Keywords: Problematic sexual behavior; Child treatment/intervention

STUDY DESIGN:
Intervention Model Description: Two conditions will be employed, PBT and treatment-as-usual, and participants will be randomly assigned to condition using a blocked randomization procedure balancing for gender and age.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of whether they are assigned to the experimental or control condition. Research assistants collecting data will similarly be unaware of the participant's condition during assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): The experimental treatment is Phase-Based Treatment (PBT) for Problematic Sexual Behavior of Preteen Children, an innovative intervention demonstrating promise in preliminary testing.
  Interventions: Behavioral: Phase-based Treatment (PBT) for Problematic Sexual Behavior of Preteen Children
- Control Treatment (Active Comparator): The Control Treatment will utilize a Treatment-as-Usual (TAU) condition designed to mimic the types of treatment generally provided in the community for mental health concerns of children.
  Interventions: Behavioral: Treatment-as-Usual (TAU)

INTERVENTIONS:
Behavioral: Phase-based Treatment (PBT) for Problematic Sexual Behavior of Preteen Children — PBT is a skills-based protocol that primarily works with caregivers to manage problematic behavior and to teach children healthy information about sex and sexuality. It was designed based on the current empirical knowledge regarding the etiology and treatment of childhood problematic sexual behavior. It is delivered in 12 weekly sessions, with each session lasting approximately 50 minutes.
  Arms: Experimental Treatment
Behavioral: Treatment-as-Usual (TAU) — The TAU intervention designed for this trial relies largely on the delivery of child-focused treatment techniques, particularly on the development of therapeutic rapport through the utilization of non-directive techniques. These sessions are supplemented with educational materials for the caregiver on child behavior and parenting recommendations. This treatment is designed to be administered over 12 weekly sessions, with each session lasting approximately 50 minutes.
  Arms: Control Treatment

SUMMARY:
Relatively little is known about the treatment of problematic sexual behavior (PSB) displayed by preteen children. Randomized controlled trials (RCTs) examining potential treatments are rare and the available results to date are generally underwhelming. A new protocol, termed Phase-Based Treatment (PBT) for Preteen PSB, has shown positive results in an early stage pilot and during community implementation efforts. This trial will be the first RCT of PBT and aim to determine whether PBT might outperform a treatment-as-usual condition.

DETAILED DESCRIPTION:
In 2015, a new intervention, PBT, was designed that relied on the current etiological research on PSB and the state-of-the-science regarding behavior change among children. A small pilot of the protocol yielded positive results. Although the pilot included only 10 participants, statistically significant pre-post changes were observed for general PSB, intrusive forms of sexual behavior, and social modeling of sexuality in the home. Training in PBT was provided to a limited number of practicing clinicians in the state of Texas and program evaluation metrics were included. Pre-post change for general PSB was significant, as were changes for intrusive forms of sexual behavior.

Despite positive outcomes in non-controlled research, it is unclear whether PBT achieves effects larger than might be seen with more general, non-specific forms of intervention. To demonstrate such an effect requires the completion of a randomized controlled trial (RCT). However, a number of feasibility issues must be answered before conducting a large scale, definitive RCT. As such, the current RCT is conceived as a feasibility project to determine the likelihood of successfully recruiting and retaining a sufficient number of participants, to derive comparative effect size estimates between PBT and SAU to inform later power analyses, and to ascertain participant satisfaction with PBT.

ELIGIBILITY:
Inclusion Criteria:

* Child between ages 4 and 12 years
* Caregiver reports a raw score on the CSBI greater than 4.
* A primary caregiver is willing to participate in treatment.
* Child earns a scaled score above 69 on the Kaufman Brief Intelligence Test (KBIT-2)
* Child proficient in spoken English
* Caregiver proficient in written and spoken English.

Exclusion Criteria:

* Child is less than 4 years of age or older than 12 years of age.
* Caregiver reports a score on the CSBI lower than 4
* A primary caregiver is unwilling to participate in treatment.
* Child scored lower than 70 on the KBIT-2.
* The primary caregiver is suspected of perpetrating child sexual abuse.
* Child not proficient in spoken English.
* Caregiver not proficient in both written and spoken English.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the Child Sexual Behavior Inventory (CSBI) | Through study completion, typically 12 weeks.
  The CSBI is a widely-used measure of problematic sexual behavior among preteen children. It is completed by caregivers and asks the frequency with which 38 different items were observed over the past six months. Caregivers report frequency using a 4-point Likert-type scale ranging from 0 (Not at all) to 3 (at least once per week).

SECONDARY OUTCOMES:
Change in scores on the Sexual Concerns subscale of the Trauma Symptom Checklist for Young Children (TSCYC) | Through study completion, typically 12 weeks.
  The TSCYC is a widely-used measure of various forms of emotional and behavioral concerns that are commonly associated with the experience of a traumatic event. One subscale, Sexual Concerns, assesses the child's display of sexual behaviors and anxiety around sexual topics. Scores are reported in T-scores, which have an average of 50 and a standard deviation of 10. Higher scores indicate greater concerns.
Change in scores on the Family Sexuality Index (FSI). | Through study completion, typically 12 weeks.
  The FSI assesses the frequency with which various forms of social modeling of sex occurs in the home. The FSI is a 14-item measure and each item is answered with a No (0) or Yes (1). The items are then summed to compute a raw score with higher scores indicating a greater display of sexuality in the home.
Change in scores on the Conduct Problems subscale of the Strengths and Difficulties Questionnaire (SDQ) | Through study completion, typically 12 weeks.
  The SDQ is a widely used measure of emotional and behavioral concerns of children. The Conduct Problems subscale specifically assessing behavioral problems, such as oppositionality, lying, and stealing. This subscale includes 5 items that are scored on a scale from 0 (Not True) to 2 (Certainly True). Higher summed scores indicate greater concerns in this area.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center-TLC Research and Treatment Center, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected data are available in a de-identified form to other researchers pending presentation of an approved IRB protocol and completion of an appropriate data usage agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available approximately 12 months after the completion of data collection.
Access Criteria: Contact the principal investigator for more information.

REFERENCES:
- [Background] Allen, B., Berliner, L., Shenk, C. E., Bendixsen, B., Zellhoefer, A., Dickmann, C. R., Arnold, B., & Chen, M. J. (2018). Development and pilot testing of a phase-based treatment for preteen children with problematic sexual behavior. Evidence-based Practice in Child and Adolescent Mental Health, 3, 274-285.
- [Background] Dickmann, C. R., Zellhoefer, A., Arnold, B., & Allen, B. (2018). Implementing a phase-based treatment for preteen children with problematic sexual behavior: Case examples. Evidence-based Practice in Child and Adolescent Mental Health, 3, 286-293.